CLINICAL TRIAL: NCT04082910
Title: Metoprolol for the Treatment of Cytokine Release Syndrome in Patients Treated With Chimeric Antigen Receptor T Cells
Brief Title: Metoprolol Treatment for Cytokine Release Syndrome in Patients Treated With Chimeric Antigen Receptor T Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-044
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Hematological Malignancy
Keywords: Metoprolol; cytokine release syndrome; chimeric antigen receptor T cells
MeSH Terms: conditions — Hematologic Neoplasms; Cytokine Release Syndrome | interventions — Metoprolol; Infliximab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conditional therapy mode group (Experimental): Metoprolol (12.5-25 mg per dose, every 12 hours) was initially given from the day of CRS diagnosis confirmation post CAR T cell infusions till CRS remission in patients without bulky tumor burden. For all metoprolol-treated patients, the use of antibodies (infliximab, etanercept and tocilizumab) and/or other agents were not completely limited under the consideration of clinical requirement for sufficient control of continuously progressed CRS.
  Interventions: Drug: Metoprolol; Drug: metoprolol, infliximab, etanercept, tocilizumab and/or other agents
- Prophylactic therapy mode group (Experimental): Metoprolol (12.5-25 mg per dose, every 12 hours) was given starting from the day before CAR T infusion till CRS remission in patients with bulky disease. For all metoprolol-treated patients, the use of antibodies (infliximab, etanercept and tocilizumab) and/or other agents were not completely limited under the consideration of clinical requirement for sufficient control of continuously progressed CRS.
  Interventions: Drug: Metoprolol; Drug: metoprolol, infliximab, etanercept, tocilizumab and/or other agents

INTERVENTIONS:
Drug: Metoprolol — Metoprolol was given in patients who received CAR T cell therapy for CRS control or CRS precaution.
Drug: metoprolol, infliximab, etanercept, tocilizumab and/or other agents — During the term of metoprolol use, antibodies (infliximab, etanercept and tocilizumab) and/or other agents were not completely limited to be used under the consideration of clinical requirement for sufficient control of continuously progressed CRS.

SUMMARY:
The aim of this prospective study is to evaluate the feasibility and efficacy of metoprolol, a beta-1 adrenergic receptor blocker, in the treatment of cytokine release syndrome (CRS) caused by chimeric antigen receptor T (CAR T) cell infusions, its effects on the serum levels of Interleukin-6 (IL-6) and other cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma, leukemia or other malignant diseases who were enrolled for CAR T cell therapy.

Exclusion Criteria:

Patients with contraindications indicated in metoprolol instruction, including:

* Significant bradycardia (heart rate < 45/min)
* Cardiogenic shock
* Severe or acute heart failure
* Poor peripheral circulation perfusion
* Grade II or III atrioventricular block
* Sick sinus syndrome
* Severe peripheral vascular disease

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of metoprolol in patients treated by CAR T infusions. | 2-4 weeks
  Reduction of heart rate in bpm (beats per minute)
Safety and tolerability of metoprolol in patients treated by CAR T infusions. | 2-4 weeks
  Reduction of blood pressure in mmHg

SECONDARY OUTCOMES:
Efficacy of metoprolol for CRS control | 2-4 weeks
  Reduction of Body temperature in degree centigrade
Efficacy of metoprolol for CRS precaution | 2-4 weeks
  Reduction of serum IL-6 in pg/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No